CLINICAL TRIAL: NCT01060735
Title: The Effect of Different Doses of Vitamin D Supplementation During Pregnancy on Bone and Vitamin D Status in Children at Birth and at One Year Age
Brief Title: Vitamin D Supplementation During Pregnancy and Bone Status in Children at Birth and at One Year of Age
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Corina Hartman, MD, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rmc005437ctil
Record Dates: First submitted 2010-01-31; First posted 2010-02-02 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Healthy
Keywords: Vitamin D; pregnancy; children; bone; quantitative ultrasound; Healthy pregnant women
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Larger doses of vitamin D supplementation (Experimental): The subjects enrolled in this arm will be supplemented during the third trimester of pregnancy with 2000IU vitamin D per day
  Interventions: Dietary Supplement: Vitamin D
- Conventional vitamin D supplementation (No Intervention): Regular supplementation during pregnancy with 400IU vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — Vitamin D 2000iu/ day from the 27 week of pregnancy up to delivery
  Arms: Larger doses of vitamin D supplementation

SUMMARY:
Vitamin D deficiency is frequently reported in pregnant women despite recommendation of daily vitamin D supplementation of 400IU/d. Recent studies have shown that in the absence of sun exposure these doses are seldom able to achieve 25(OH)D optimal serum levels.

We hypothesize that larger doses of vitamin D are needed to be supplemented to all women during pregnancy. We hypothesize that this may have advantageous effects on maternal vitamin D and bone reserve as well on offspring vitamin D and bone status at birth and possible further on.

The aim of the present study is to compare vitamin D and bone status of infants born to mothers supplemented with 400IU/d (present recommendations) and 2000IU/d vitamin D during the third trimester of pregnancy.

DETAILED DESCRIPTION:
This is a prospective randomized controlled study.

120 pregnant women will be recruited at 27 weeks gestation and randomized into two treatment groups; 400IU/d or 2000IU/d vitamin D supplementation from 27 weeks until delivery.

25-hydroxyvitamin D (25OHD), parathyroid hormone (PTH), urinary calcium/creatinine and serum calcium and alkaline phosphatase (ALP) levels will be assessed in mothers at 27 weeks and at delivery.

25OHD, calcium and ALP levels, and urinary calcium/creatinine will be evaluated in offspring at birth and at one year age.

Vitamin D and calcium intake and sun exposure will be evaluated in mothers and offsprings.

Quantitative ultrasound (QUS) measurement of tibia and radius will be performed to newborns and at the age of one year.

Bone status of newborns at birth and at one year age in children will be compared between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women aged 20 to 40 years, of any parity status.
* Signed informed consent

Exclusion Criteria:

* Presence of diseases known to affect vitamin D status such as malabsorption states, liver and renal disorders, primary and tertiary hyperparathyroidism, granulomatous disorders
* Treatment with medications known to affect vitamin D status such as anticonvulsivants, glucocorticoids, antirejection medication and retroviral agents

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Bone status in offspring at the age of one year as assessed by tibial and radius quantitative ultrasound (QUS). | Bone status in offsprings, assessed at the age of one year

SECONDARY OUTCOMES:
Vitamin D status of mothers. | At the start of intervention, at delivery and at the age of one year
Maternal health status. | At the start of intervention, at delivery and at the age of one year
Infants' growth. | At the start of intervention, at delivery and at the age of one year
Vitamin D status in infants. | At the start of intervention, at delivery and at the age of one year
Safety of vitamin D supplementation doses. | At the start of intervention, at delivery and at the age of one year

CONTACTS AND LOCATIONS:
Overall Officials: Corina Hartman, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel